CLINICAL TRIAL: NCT05258721
Title: Efficacy of ClōSYS® Sensitive Fluoride Toothpaste and ClōSYS® Sensitive Rinse Regimen on Plaque, Gingival Inflammation and Bleeding Upon Probing
Brief Title: Efficacy of ClōSYS® Sensitive Fluoride Toothpaste and ClōSYS® Sensitive Rinse Regimen on MGI, PI and BOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rowpar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATSU-RPR-Oral rinse 2020
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Gingivitis; Periodontitis
Keywords: Gingivitis or periodontitis (Stage I or II)
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Participants with gingivitis or periodontitis (Stage I or II) brush with ClōSYS® Sensitive Fluoride Toothpaste twice daily and rinse with ClōSYS® Sensitive Rinse twice daily after brushing.
  Interventions: Drug: ClōSYS® Sensitive Fluoride Toothpaste; Other: ClōSYS® Sensitive Rinse

INTERVENTIONS:
Drug: ClōSYS® Sensitive Fluoride Toothpaste — ClōSYS® Sensitive Fluoride Toothpaste is an over-the-counter drug product containing 0.12% stabilized chlorine dioxide (sodium chlorite in an aqueous solution) and 0.13% w/v fluoride ion.
Other: ClōSYS® Sensitive Rinse — ClōSYS® Sensitive Rinse is a cosmetic product containing 0.1% stabilized chlorine dioxide.

SUMMARY:
90-day, self-controlled, longitudinal, non-blinded clinical trial which will measure changes in clinical parameters in participants with gingivitis and Stage I or II periodontitis who apply ClōSYS® Sensitive Fluoride Toothpaste and ClōSYS® Sensitive Rinse.

DETAILED DESCRIPTION:
The study will be conducted with 60 medically healthy participants between ages 18 to 75 years with gingival or periodontitis (Stage I or II) who are receiving routine preventive care and/or periodontal maintenance.

Subjects will brush with ClōSYS® Sensitive Fluoride Toothpaste twice daily and rinse with ClōSYS® Sensitive Rinse twice daily after brushing.

The primary response variables will be the Subjects' scores on the Plaque Index (PI), Gingival Index (GI) and the number of sites with bleeding upon probing (BOP). Probing depths and clinical attachment level will be assessed at baseline and 3 months. Adverse events will also be assessed and documented at each visit. In addition, Subjects will keep a usage diary documenting their daily use of the toothpaste and oral rinse and any comments or observations regarding usage or adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between the ages of 18 to 80 years
* Subjects have a minimum of 20 permanent teeth, excluding third molars
* Subjects have been diagnosed with gingivitis or periodontitis (Stages I and II are based on the level of CAL and Bone Loss (BL). The diagnosis is Stage I if: (a) BL is less than 15% and (b) CAL is between 1-2mm. The diagnosis is Stage II if: (a) BL is between 15% and 33% and (b) CAL is between 3-4mm)
* Subjects exhibit bleeding upon probing in >20% of sites
* Subject is seen every 3 months for routine dental prophylaxis/periodontal maintenance
* Subjects do not have a significant medical history or metabolic diseases (diabetes with A1C ≥ 7.0, pregnancy)
* Subject is currently a non-smoker or has discontinued smoking at least 6 months prior to enrollment
* Subject agrees to refrain from use of the following products: Peridex®, PerioGuard®, Listerine®, Cepacol®, Crest Pro-Health® rinse, Colgate Total® rinse, Colgate Total® toothpaste, Crest Pro Health® toothpaste, or any generic equivalent while participating in this study. Alcohol is not the active ingredient in any oral rinse product and does not produce a significant antibacterial effect
* Subject is able to read and provide written informed consent
* Subject is able to follow verbal and/or written instructions, perform oral hygiene procedures and return to the test facility for specified study examinations
* Subject agrees not to receive a dental "cleaning" (prophylaxis) while in the study
* Subject must permanently reside in Arizona

Exclusion Criteria:

* Subject has significant medical history or poorly controlled/uncontrolled diabetes (as defined above)
* Subject is pregnant
* Subject has a medical condition that requires antibiotic premedication prior to dental treatment
* Subject has taken antibiotics within 1 month of study enrollment
* Subject who takes multiple medications and/or herbal and dietary supplements known to alter bleeding and exhibits/reports spontaneous gingival bleeding
* Subject takes medications that may interfere with study results (eg. antibiotics, steroids, immunosuppressants, high dose aspirin (325+ mg/day), chemotherapy and/or radiation therapy for cancer).
* Subject is a current smoker
* Subject has a history of non-surgical or surgical periodontal therapy within 6 months of study participation
* Subject has Stage III or IV periodontitis, Grade B or C
* Subject is currently taking or in the past 28 days has taken another investigational drug or participated in other investigational studies that may impact study outcomes
* Subject has not had a dental cleaning within six months prior to the start of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaiprakash Shewale, Ph.D., Study Director — Rowpar Pharmaceuticals, Inc.
Locations (1):
- Arizona School of Dentistry & Oral Health, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 60
Completed | 52
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Modified Gingival Index (MGI)
Description: MGI uses a rating score between 0 and 4, with 0 indicating a tooth with healthy gums and 4 the most severe inflammation. MGI scores were determined by visual exam of the gingiva on 4 surfaces for each tooth present except for third molars, for a total of 28 teeth. The total number of teeth exhibiting inflammation affecting all portions of the gingival unit (Score ≥ 2) were noted at each visit. The total number of teeth affected was evaluated for each visit in the final analysis.
  At baseline: Score range is (0-64) At 12 weeks: Score range is (0-32)
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 52
score on a scale
  Baseline | 8.5 [4.0 to 16.25]
  12 weeks | 1.5 [0.0 to 4.25]
Statistical Analysis 1: Comparison: Treatment Group; Test type: Superiority; p < 0.001, Kruskal-Wallis

2. Primary Outcome: Changes in Plaque Index (PI)
Description: The PI was recorded on all teeth except for third molars. PI was recorded on 4 surfaces of each tooth. PI uses a rating score between 0 and 3, with 0 indicating no plaque in gingival area and 3 heavy accumulation of plaque. Total score is reported.
  At baseline: Score range is 9 -157. At 12 weeks: Score range is 1 -147.
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 52
score on a scale
  Baseline | 22.0 [15.0 to 40.0]
  12 weeks | 8.0 [5.75 to 17.5]
Statistical Analysis 1: Comparison: Treatment Group; Test type: Superiority; p < 0.001, Kruskal-Wallis — The threshold for statistical significance was p =0.05

3. Primary Outcome: Changes in Bleeding On Probing (BOP)
Description: Bleeding On Probing (BOP) will be recorded as a dichotomous variable (present/absent) during the periodontal examination. The percentage of sites that bleed will be calculated by dividing the number of sites with bleeding by the total number of sites.
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of sites with bleeding
Arm/Group | Treatment Group
Number analyzed (Participants) | 52
percentage of sites with bleeding
  Baseline | 37.0 [29.0 to 45.0]
  12 weeks | 15.0 [10.0 to 24.25]
Statistical Analysis 1: Comparison: Treatment Group; Test type: Superiority; p < 0.001, Wilcoxon signed rank test

4. Secondary Outcome: Adverse Events
Description: Adverse events will be collected throughout the study
Time Frame: 90 Days
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 52
participants | 0

ADVERSE EVENTS:
Time Frame: From Baseline Visit 1 to End of the study Visit 3 (12 weeks/3 months)
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT05258721/Prot_SAP_001.pdf